CLINICAL TRIAL: NCT02922738
Title: The Impact of a Dermatology Information Source on Skin Problem Outcomes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Marianne Burke, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHRMS 15-413
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Decision Support Systems,Clinical; Skin Diseases
Keywords: Clinical Knowledge Systems, Decision support, Dermatology; Technology Assessment
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - VisualDx Arm (Experimental): Arm had 2 levels: provider (cluster) level and patient level. Providers, randomly assigned to the intervention arm, refer to VisualDx when they saw a patient who presented with a skin problem. Their patients were assigned to the intervention group and interviewed about the outcomes of their treatment.
  Interventions: Other: VisualDx
- Control - Usual Care Arm (No Intervention): Arm had 2 levels: provider (cluster) level and patient level. Providers, randomly assigned to control, did not refer to VisualDx but could refer to other information sources or none per usual care. Their patients were assigned to the control group and interviewed about the outcomes of their treatment

INTERVENTIONS:
Other: VisualDx — VisualDx is a computerized clinical information technology with medical image and text content in dermatology.
  Arms: Intervention - VisualDx Arm

SUMMARY:
Health care providers use a variety of computerized medical information sources to reduce knowledge gaps and support patient care decisions. Few studies have evaluated the impact of medical information sources on patient outcomes. Skin problems are the reason for many visits to primary care providers and result in a high percentage of referrals to dermatologists and return visits to primary care for the same skin problem.

The objective is to evaluate the impact of primary care providers' use of a dermatology information source, VisualDx, on skin problems outcomes.

The study design is a cluster-randomized controlled trial. Participants include primary care providers as clusters and their patients with skin problems. Providers are randomized to intervention group that refers to VisualDx when seeing a patient with a skin problem, or to the control group who does not. Patients have the randomized group status of the doctor they saw for the problem.

Patients are interviewed to determine the problem status and how many follow-up visits they had for the problem at intervals after the index visit.

DETAILED DESCRIPTION:
The research design is a cluster randomized controlled trial of a computerized dermatology information source. This is a two-level design in which primary care providers (PCPs) who see patients for skin problems are the subjects of randomization. Their patients are the subjects of the data collection and analysis. The cluster design examines how much variation in the outcomes is attributable to the providers, how much to patients within the clusters, and how much to the intervention information source itself.

Provider Level:

After completing a baseline questionnaire, providers are randomized to intervention or control groups. Intervention group providers have an orientation to the study protocol that includes how to access and use VisualDx. Control providers receive the protocol overview, but no orientation to the intervention.

Intervention providers agree to refer to VisualDx content when they have a patient with a skin complaint. Control group providers agree not use VisualDx as a reference but may use another medical information source or none.

Patient Level:

To identify eligible patients, authorized investigators reviewed information from the patient record sufficient to send a letter to them over the provider's signature to notify them about the study. The letter gives the option to refuse any contact.

At 30 days after the primary care visit, a study team investigator phones each eligible patients, explains the study, and obtains verbal consent. The investigators are blinded to the randomized group status of the patients.

The investigator proceeds with the interview questionnaire on consent. Age, sex is collected. Patients are asked whether the skin problem is resolved ("Is it all better?"). For every resolved problem, we ask when (date or days since visit) it was resolved. We also ask how many return visits the patient has had with any provider for that problem.

If not resolved, the patient is called again at 60 days and asked the same questions. If not resolved then, we call the patient again at 90 days. The last call to any patient is at 90 days from the index visit for the problem.

Data Analysis and Statistical Measures

The primary predictor variable for both aims is the use of the VisualDx information source by the primary care provider.

For the "days to resolution" outcome variable, the time unit (days) and the status of the problem after 90 days (resolved or not resolved) will be evaluated for each group with Kaplan-Meier survival analysis and the non-parametric log rank test of significance.

For the "number of follow-up visits" outcome variable, the binary predictor (intervention group) and discrete outcome variable (number of visits) will be evaluated with Wilcoxon-rank sum test for non-normal data. The first visit of a patient to a participating provider for a skin problem is considered the index visit and that provider considered the index provider regardless of the provider seen on any subsequent appointment. Analysis will adhere to the intention-to-treat principle with group assignment determined by randomization regardless of whether VisualDx was deployed for care or not. Problems unresolved at the last contact will be censored as unresolved for the Kaplan-Meier analysis.

For aim 1, the estimated sample size to detect an average difference of 8 days in time to resolution with a standard deviation of 20 and an intra-cluster correlation (ICC) of 0.025. With alpha .05 and beta .80, the study would need a minimum 26 providers enrolled with an average 10 patient participants in each provider's cluster for a total of 286 participants completing the study. We planned to enroll at least 30 providers and up to 500 patients to insure against loss to follow-up of, increased standard deviation, or larger than anticipated Intra-Cluster Correlation.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by a participating Primary Care Provider for a chronic or acute skin problem

Exclusion Criteria:

* Skin problems due to burns or lacerations
* Cognitively impaired, mentally ill, prisoners, non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne D Burke, PhD, Principal Investigator — University of Vermont; Benjamin Littenberg, MD, Study Chair — University of Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alper BS, White DS, Ge B. Physicians answer more clinical questions and change clinical decisions more often with synthesized evidence: a randomized trial in primary care. Ann Fam Med. 2005 Nov-Dec;3(6):507-13. doi: 10.1370/afm.370. PMID 16338914
- [Background] Del Fiol G, Haug PJ, Cimino JJ, Narus SP, Norlin C, Mitchell JA. Effectiveness of topic-specific infobuttons: a randomized controlled trial. J Am Med Inform Assoc. 2008 Nov-Dec;15(6):752-9. doi: 10.1197/jamia.M2725. Epub 2008 Aug 28. PMID 18755999
- [Background] Marshall JG, Sollenberger J, Easterby-Gannett S, Morgan LK, Klem ML, Cavanaugh SK, Oliver KB, Thompson CA, Romanosky N, Hunter S. The value of library and information services in patient care: results of a multisite study. J Med Libr Assoc. 2013 Jan;101(1):38-46. doi: 10.3163/1536-5050.101.1.007. PMID 23418404
- [Background] Isaac T, Zheng J, Jha A. Use of UpToDate and outcomes in US hospitals. J Hosp Med. 2012 Feb;7(2):85-90. doi: 10.1002/jhm.944. Epub 2011 Nov 16. PMID 22095750
- [Background] Awadalla F, Rosenbaum DA, Camacho F, Fleischer AB Jr, Feldman SR. Dermatologic disease in family medicine. Fam Med. 2008 Jul-Aug;40(7):507-11. PMID 18928078
- [Background] Federman DG, Reid M, Feldman SR, Greenhoe J, Kirsner RS. The primary care provider and the care of skin disease: the patient's perspective. Arch Dermatol. 2001 Jan;137(1):25-9. doi: 10.1001/archderm.137.1.25. PMID 11176657
- See also: VisualDx [Internet]. Logical Images, Inc. . Available by individual and institutional license. — https://www.visualdx.com/visualdx/7/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Provider recruitment by email invitation to Family Medicine and Adult Medicine providers at one academic medical center. 32 primary care providers (PCPs) enrolled. 989 patients with a skin problem visit to a participating PCP were identified between November 2015 to August, 2016. 433 patients participated by providing data in telephone interviews.
Groups:
- Intervention - VisualDx Arm: Providers (clusters) randomized to use VisualDx when seeing a patient that presented with a skin problem. Their patients, seen for a skin problem were interviewed for outcome data.
- Control: Usual Care Arm: Control providers (clusters) did not use VisualDx but could refer to other information sources or none in usual care.
Period: Overall Study
Arm/Group | Intervention - VisualDx Arm | Control: Usual Care Arm
Started | 175 (158 patients and 17 providers) | 290 (275 patients and 15 providers)
Completed | 175 | 290
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention - VisualDx Arm: Providers referred to VisualDx when seeing a patient with a skin problem. Patients with skin problem were interviewed for outcomes data.
- Control - Usual Care Arm: Providers ddi not refer to VisualDx but could refer to other resources or none per usual care.
- Total: Total of all reporting groups
Arm/Group | Intervention - VisualDx Arm | Control - Usual Care Arm | Total
Number analyzed (Participants) | 175 | 290 | 465
Age, Continuous [Median (Full Range); unit: years] — Age data were collected for patients only. Population: Age data were collected for patients only.
  years
    number analyzed (Participants) | 158 | 275 | 433
    (all) | 58 [20 to 91] | 58 [19 to 94] | 58 [19 to 94]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex measure includes both provider participants and patient participants. 2 patients, 1 intervention and 1 control, did not provider sex data. Population: 2 patients, 1 intervention and 1 control, did not provide sex data.
  Participants
    Patients: number analyzed (Participants) | 157 | 274 | 431
    Patients: Female | 80 | 137 | 217
    Patients: Male | 77 | 137 | 214
    Providers: number analyzed (Participants) | 17 | 15 | 32
    Providers: Female | 7 | 8 | 15
    Providers: Male | 10 | 7 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 175 | 290 | 465

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Resolved Skin Problems
Description: Resolved skin disease status was assessed by phone interview. Patient reported status. Patients were censored if "unresolved" at 90 days.
Time Frame: Period of assessment was up to 3 months (90 days) after index visit.
Population: Number of patient participants only (excludes providers)
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Used VisualDx: Providers referred to VisualDx when seeing a patient that presented with a skin problem. Patients were interviewed about the outcome of their treatment. Patients were allocated to the randomization group of the PCP they saw.
  VisualDx: VisualDx is a computerized clinical information technology with medical image and text content in dermatology.
- Control - Usual Care: Providers did not use VisualDx but may have referred to other information sources or none (usual care). Patients were allocated to the randomization group of the PCP they saw.Patients were interviewed about the outcome of their treatment.
Arm/Group | Intervention - Used VisualDx | Control - Usual Care
Number analyzed (Participants) | 158 | 275
Participants | 72 | 135
Statistical Analysis 1: Comparison: Intervention - Used VisualDx vs Control - Usual Care; Test type: Superiority; p = 0.54, Regression, Cox; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.70 to 1.21]

2. Primary Outcome: Number of Follow-Up Visits to Any Provider for the Same Problem
Description: Follow-up visits count is assessed at each phone interview. Patients report return visits.
Time Frame: Period of Assessment is up to 90 days after index visit
Measure: Median (Full Range); unit: Return Appointments
Groups:
- Intervention - Used VisualDx: Providers referred to VisualDx when seeing a patient that presented with a skin problem. Patients were interviewed about the outcome of their treatment. Patients were allocated to the randomization group of the PCP they saw.
  VisualDx: VisualDx is a computerized clinical information technology with medical image and text content in dermatology.
  Providers were the subjects of randomization. Patients were the subjects of analysis.
- Control - Usual Care: Providers did not use VisualDx but may have referred to other information sources or none (usual care). Patients were allocated to the randomization group of the PCP they saw.Patients were interviewed about the outcome of their treatment.
  Providers were the subjects of randomization. Patients were the subjects of analysis.
Arm/Group | Intervention - Used VisualDx | Control - Usual Care
Number analyzed (Participants) | 158 | 275
Return Appointments | 0.65 [0 to 7] | 0.55 [0 to 7]
Statistical Analysis 1: Comparison: Intervention - Used VisualDx vs Control - Usual Care; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring began on recruitment of provider participants through completion of patient interviews: August 2015 through October 2016, approximately 14 months.
Description: We hypothesized that there were minimal risks to participants such as loss of time spent learning new information or answering questions by providers and loss of privacy by patients, but protected health information was only exposed to treating physicians, the Principal Investigator and study team. Other hypothesized minimal patient risks included the bother of phone calls and loss of time spent answering questions. Adverse events were monitored for both patient and provider participants.
Groups:
- Intervention - Used VisualDx: Providers referred to VisualDx when seeing a patient that presented with a skin problem. Patients were interviewed about the outcome of their treatment. Patients were allocated to the randomization group of the PCP they saw.
  VisualDx: VisualDx is a computerized clinical information technology with medical image and text content in dermatology.
  Providers were the subjects of randomization. Patients were the subjects of analysis.
  There were no adverse events reported.
- Control - Usual Care: Providers did not use VisualDx but may have referred to other information sources or none (usual care). Patients were allocated to the randomization group of the PCP they saw.Patients were interviewed about the outcome of their treatment.
  Providers were the subjects of randomization. Patients were the subjects of analysis.
  There were no adverse events reported.
Arm/Group | Intervention - Used VisualDx | Control - Usual Care
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/290
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/290
Other Adverse Events (participants affected / at risk) | 0/175 | 0/290

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No